CLINICAL TRIAL: NCT04037215
Title: Exploration of the Mechanisms of Vulnerability of Anorexia Nervosa at an Early Age : Study of the Cognitive Treatment of Food Stimuli and Body Image
Acronym: AMDP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: K170607J
Record Dates: First submitted 2019-07-26; First posted 2019-07-30 (Actual); Last update posted 2021-10-18 (Actual); Status verified 2021-10

CONDITIONS: Anorexia Nervosa
Keywords: eye tracking; cognitive processing
MeSH Terms: conditions — Anorexia Nervosa

STUDY DESIGN:
Intervention Model Description: All assessments in patients with AM are performed as part of routine care and do not require additional monitoring modalities added by research.
  For controls, phenotypic exploration will require a consultation with clinical examination including the search for psychiatric comorbidities and the completion of standardized questionnaires, exploration of the neuropsychological profile (with eye tracking, overall cognitive exploration, executive functions, social cognition and self-esteem).
  Test results will not be returned except for screening requiring specific management. The information will then be returned to the child's parents by the investigating doctor, who will be responsible for organizing specific care whenever it is necessary.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- COGNITIVE TREATMENT OF DIETARY STIMULI AND BODY IMAGE (Other): In order to explore the cognitive treatment of patients with early onset anorexia nervosa in front of images of silhouettes and food, it is currently used in the child psychiatry department of the Robert Debré Hospital, the eye-tracking method. Eye tracking is a non-invasive and painless method of recording the path of vision on images presented on a computer screen. In order to understand the specificities of the eye path in sick patients, we will compare the data with those of controls without eating disorders.
  Interventions: Other: STUDY OF THE COGNITIVE TREATMENT OF DIETARY STIMULI AND BODY IMAGE

INTERVENTIONS:
Other: STUDY OF THE COGNITIVE TREATMENT OF DIETARY STIMULI AND BODY IMAGE — Describe the cognitive treatment of patients with early onset anorexia nervosa in response to specific stimuli of the disorder (eating and body images), compared to age- and sex-matched control subjects:
  * children controls not achieved with normal BMI;
  * children with unbalanced insulin-dependent type 1 diabetes, therefore subject to a strict diet that requires good nutritional knowledge and no weight judgment disorders.

SUMMARY:
In order to explore the cognitive treatment of patients with early onset anorexia nervosa (AM) in front of images of silhouettes and food, we will use the eye-tracking method. While we hypothesize a judgment disorder in these patients, the exploration of implicit cognitive treatment without desirability bias is essential. Eye-tracking is a method of recording the eye path that provides qualitative and quantitative information on the visual exploration of subjects. The visual pathway depends on how the subject's attention is directed to a given stimulus, but also on certain cognitive traits (e.g., excessive attention to details) or symptoms (e.g., avoidance of caloric food images or attraction to thin images). It is therefore a non-invasive exploration tool, which provides information on how patients look at food images and silhouettes. This project will describe the cognitive treatment of dietary stimuli and body image in young patients with early onset AM. It could identify a biomarker of AM in the pediatric population and improve the diagnosis of the disease. A better diagnosis of AM in patients under 15 years of age is essential and will improve medical care and develop personalized medicine.

DETAILED DESCRIPTION:
Monocentric, prospective cohort, case-control type study. The population concerned is composed of patients with early onset anorexia nervosa (AM) and control subjects (two groups).

The objectives of this study are to:

Describe the cognitive treatment of early-onset AM patients with specific stimuli of the disorder (eating and body images) compared to age- and sex-matched control subjects:

* children controls not achieved with normal body mass index(BMI);
* children with unbalanced insulin-dependent type 1 diabetes, therefore subject to a strict diet that requires good nutritional knowledge and no weight judgment disorders.

Describe the links between cognitive treatment and clinical phenotype in patients with early onset AM, in particular severity of eating behaviour trouble symptomatology (TCA), psychiatric and somatic comorbidities, neuropsychological profile.

30 patients with early-onset AM. Two groups of control subjects (matched for age and gender): 30 subjects from the general population with a normal Body Mass Index (BMI) and 30 subjects with chronic somatic pathology (type 1 diabetes) without weight variation (good knowledge of dietary caloric values without impaired judgment about the caloric value of foods and representation of the body image of self and others) A total of 90 participantsPatients and controls without eating disorders will be recruited at Robert Debré Hospital, after signature of the authorization by the holder(s) of parental authority present at the time of hospitalization All patients treated in the department benefit from extensive phenotypic exploration, carried out in routine care.

For controls, phenotypic exploration will require a half-day evaluation.

ELIGIBILITY:
Inclusion Criteria:

Patients with anorexia nervosa.

* Age 8 to 14 years,
* Early AM diagnosis (AM DSM-5 criteria, and presence of primary amenorrhea at diagnosis for girls),
* Follow-up in the Child Psychiatry Department of the Robert Debré Hospital,
* Affiliation to a social security system,
* Authorization of the holder(s) of parental authority and acceptance of the child to participate in this research.

Witnesses from the general population:

* Age 8 to 14 years,
* Normal Height-weight development defined by: Weight, Height, BMI between 10° and 90° percentile for age and sex, without changing the growth curve.
* Authorization of the holder(s) of parental authority and acceptance of the child to participate in this research

Witnesses with type 1 diabetes:

* Age 8 to 14 years,
* Type 1 diabetes for more than a year,
* Follow-up in the endocrinology department of the Robert Debré Hospital,
* Normal height-weight development defined by: Weight, Height, BMI between 10° and 90° percentile for age and sex, without changing the growth curve.
* No clear imbalance with HbA1c <8.5%.
* Authorization of the holder(s) of parental authority and acceptance of the child to participate in this research

Exclusion Criteria:

* Patients with AM.
* Existence of an intellectual deficit (IQ <70). The patient will not be able to have a new IQ test within one year of inclusion.
* Other Axis I disorder (Kiddie SAS)
* Existence of a severe neurosensory disorder
* Existence of a neurological disorder
* other eating disorders(DSM-5)
* Diabetes type 1

Witnesses :

* Any Axis I psychiatric disorder
* Existence of an intellectual deficit
* Existence of a severe neurosensory disorder
* Existence of a neurological disorder
* Long-term drug treatment (other than insulin for controls with type 1 diabetes)
* Type 1 diabetes (for controls in the general population)

Psychometric test taken in the year before inclusion

Ages: 8 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Estimated)
Dates: Start 2019-11-19 (Actual); Primary Completion 2022-12-19 (Estimated); Study Completion 2022-12-19 (Estimated)

PRIMARY OUTCOMES:
cognitive processing | one day
  cognitive processing in front of 20 images of food and silhouettes of variable weight

SECONDARY OUTCOMES:
fixing a region of interest | one day
  Variables on Eye Tracking ,presence or not of a fixation of a region of interest is defined as a stabilized look at an area of 30 pixels radius for at least 100ms
body mass index | one day
  severity of symptomatology of the eating disorder
total score on the Morgan and Russell scale | one day
  severity of symptomatology of the eating disorder. Morgan and Russell's (or Global Outcome Assessment Scale), MRS (Morgan and Hayward 1988). Morgan and Russell scales are used to assess the main aspects of anorexia nervosa

CONTACTS AND LOCATIONS:
Overall Officials: Clarke Julia, PhD, Principal Investigator — APHP
Locations (1):
- Hôpital Robert Debré, Paris, France